CLINICAL TRIAL: NCT02996422
Title: Appalachians Together Restoring the Eating Environment (Appal-TREE): Advancing Sustainable CBPR Interventions to Improve Healthy Diet in Rural Appalachian Children
Brief Title: Appalachians Together Restoring the Eating Environment: Improving Healthy Diet in Rural Appalachian Kentucky
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Swanson, PhD (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Community Farm Alliance (Other)
Responsible Party: Sponsor-Investigator, Mark Swanson, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-0245-P3H; U01MD010556 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-19 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Feeding Behavior; Drinking Behavior
MeSH Terms: conditions — Feeding Behavior; Drinking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School-based water campaign (Experimental): Students who attend middle and high schools in the intervention counties will receive a school-based water campaign. A sample of students from each school will complete surveys before and after the installation of the water refilling stations to measure beverage consumption, knowledge, attitudes, and self-efficacy.
  Interventions: Behavioral: School-based water campaign
- Comparison schools (No Intervention): A sample of students who attend middle and high schools in the comparison county, which does not receive any intervention components, will complete surveys to measure beverage consumption, knowledge, attitudes, and self-efficacy.
- Community cooking classes (Experimental): Adults in the same intervention counties as the school-based water campaign will enroll in group cooking classes. They will complete a baseline and two follow-up surveys to measure changes in fruit and vegetable consumption, attitudes, and self-efficacy.
  Interventions: Behavioral: Community cooking classes

INTERVENTIONS:
Behavioral: School-based water campaign — Includes: 1) the installation of filtered water bottle refilling stations, 2) the distribution of reusable water bottles to all students and teachers, and 3) a social marketing campaign to support the increase of water consumption among students.
  Arms: School-based water campaign
Behavioral: Community cooking classes — Cooking classes will be delivered to groups of 8-12 adult participants as a series of 8 weekly classes in community venues. The content of each class is driven by topics and themes identified and prioritized by community members, namely cooking healthy on tight budget.
  Arms: Community cooking classes

SUMMARY:
Most of the nation's serious chronic health challenges and causes of death, including diabetes, heart disease, cancer, and obesity, are directly linked to sub-optimal diet. Both poor diets and associated disease are disproportionately common in the Appalachian counties of eastern Kentucky, a region with stark health inequities, including elevated rates of obesity, overweight, and premature mortality. The purpose of this study is to evaluate a multi-component intervention developed through community-based participatory research methods for improving access to healthy foods and enhancing dietary intake in eastern Kentucky. The intervention components evaluated in this study consist of: 1) a school-based campaign to promote water consumption in middle and high schools and 2) a series of group cooking classes for adults.

ELIGIBILITY:
Inclusion Criteria:

* For school-based component: Student in selected middle or high school classroom in a participating school in intervention or comparison counties (6th to 12th grades)
* For cooking classes: adult aged 18 years or older and residing in intervention county who have at least one dependent child attending middle or high school in the participating school districts

Exclusion Criteria:

* Unable to speak or read English, as all materials will be presented in English

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1657 (Actual)
Dates: Start 2016-11; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in beverage consumption (students) | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months
  Survey items address frequency and quantity of beverages consumed in past month. Includes water, pop/soda, diet pop/soda, sports drinks, energy drinks, sweetened tea, 100% fruit juice, and milk.
Change in fruit and vegetable consumption (adults) | Baseline to 8 weeks
  Survey items address frequency and quantity of consumption of fruits and vegetables in the past month.

SECONDARY OUTCOMES:
Change in attitudes and preferences about beverages (students) | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months
  Survey items address taste preferences, attitudes about eating/drinking behavior and body image, and self-efficacy.
Change in purchasing of drinks (students) | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months
  Survey items will address frequency of purchasing beverages at fast food restaurants, convenience stores, and school venues and events.
Change in food preparation habits (adults) | Baseline to 8 weeks
  Survey items address meal planning and preparation
Change in food purchasing habits (adults) | Baseline to 8 weeks
  Survey items address frequency of purchasing food at work, grocery/convenience stores, restaurants and produce stands
Change in perceptions of availability of health foods (adults) | Baseline to 8 weeks
  Survey items address availability of high quality fruits and vegetables and low-fat foods
Change in barriers to health eating (adults) | Baseline to 8 weeks
  Survey items address physical, psychosocial, emotional, and financial barriers to healthy eating

CONTACTS AND LOCATIONS:
Overall Officials: Mark Swanson, PhD, Principal Investigator — University of Kentucky

IPD SHARING:
Plan to Share IPD: No